CLINICAL TRIAL: NCT06248905
Title: Shock Wave Therapy Combined With Strengthening Exercise of Hip Abductor Muscles in the Greater Trochanteric Pain Syndrome: a Randomized Controlled Trial
Brief Title: Shock Wave Therapy Plus Exercise in GTPS
Acronym: GTPSSWEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Ettore Carlis, Medicine Doctor, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0005201/24
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Greater Trochanteric Pain Syndrome of Both Lower Limbs
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise plus shockwaves (Experimental): Enrolled subject will be treated with focused shock wave therapy, once a week for three consecutive weeks, by a specialized physician, using a device powered by an electromagnetic generator.
  Focusing: (out-of-line) ultrasound-guided with the patient lying in lateral decubitus.
  Dosimetry: 1500-1800 shots per session with an energy flux density equal to 0.10-0.20 mJ/mm2 (frequency=4Hz).
  The experimental group will then start a physiotherapy program for the following 8 weeks. The program is made up of strengthening and stretching exercises of gluteal muscles, planned to be daily performed at home. Four supervised physiotherapy session will be planned on week 0-1-2-4, during which the exercise loading will be implemented.
  Interventions: Other: Rehabilitation program based on the strengthening of gluteal muscles; Other: Extracorporeal shock wave therapy
- shockwaves (Active Comparator): Enrolled subject will be treated with focused shock wave therapy, once a week for three consecutive weeks, by a specialized physician, using a device powered by an electromagnetic generator.
  Focusing: (out-of-line) ultrasound-guided with the patient lying in lateral decubitus.
  Dosimetry: 1500-1800 shots per session with an energy flux density equal to 0.10-0.20 mJ/mm2 (frequency=4Hz).
  Interventions: Other: Extracorporeal shock wave therapy

INTERVENTIONS:
Other: Rehabilitation program based on the strengthening of gluteal muscles — Physiotherapy program (8 weeks)
  Arms: exercise plus shockwaves
Other: Extracorporeal shock wave therapy — Focused shock wave therapy (3 weeks)

SUMMARY:
The aim of this randomized controlled study is to investigate if the sequential administration of focused shock wave therapy and of a rehabilitation program based on the strengthening of gluteal muscles is more effective than a standard shock wave treatment for greater trochanteric pain syndrome

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hip pain of four weeks or longer duration
* Pain to palpation in the greater trochanteric area at physical examination
* Pain in hip end-range abduction/rotation/adduction at physical examination
* Gluteal tendinopathy, in absence of full thickness tears at a sonographic examination of the gluteal tendons
* Adult age and written informed consent

Exclusion Criteria:

* No hip osteoarthritis, diagnosed according to Altman's criteria
* No history of knee osteoarthritis
* No history of rheumatologic diseases
* No previous fractures or surgery in the affected limb
* No clinical signs of lumbar radiculopathy at physical examination
* No corticosteroid injections, since the onset of the current pain episode
* No general contraindication to shock wave therapy (pregnancy, bleeding disorders or anticoagulant drug usage, cancer in the focal area)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
NRS Pain | 6 months
  Change in lateral hip pain measured by the Numeric Rating Scale (NRS)

SECONDARY OUTCOMES:
EQ5D Quality of life | 12 months
  Change in quality of life measured by EQ-5D-3L
VISA-G Disability | 12 months
  Change in disability measured by VISA-G questionnaire
Functional capacity (strength of gluteal muscles) | 12 months
  Change in functional capacity measured by MRC scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy